CLINICAL TRIAL: NCT01104246
Title: An Open Label, Dose-Titration Investigation of the Pharmacokinetics, Metabolism and Safety of Testosterone Transdermal Systems in Hypogonadal Men
Brief Title: Dose Titration Investigation of the Pharmacokinetics of Testosterone Transdermal Systems in Hypogonadal Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AND1001
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone; Hormone replacement therapy
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone Transdermal Systems (Experimental): Testosterone
  Interventions: Drug: Testerone Transdermal System

INTERVENTIONS:
Drug: Testerone Transdermal System — Transdermal testosterone applied daily for 4 weeks
  Other Names: Testosterone

SUMMARY:
The study will evaluate the pharmacokinetics of testosterone transdermal systems at steady-state in hypogonadal men.

DETAILED DESCRIPTION:
Subjects will receive testosterone for 4 weeks. Based on a single morning testosterone measurement performed at the end of Week 1, the dosage can be titrated up or down to the next dose level to maintain testosterone levels in the normal range. At the end of 4 weeks of treatment, a pharmacokinetic profile for total testosterone and metabolites will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Males in good general health, 18 years of age or older.
* Have a previously documented testosterone deficiency.
* Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Have a history of intolerance to Androderm or other testosterone products.
* Prostate specific antigen (PSA) level ≥ 4.0 ng/mL
* Prostate cancer or severe benign prostatic hypertrophy (BPH)
* Have significant abnormalities in the physical examination at screening.
* Have current dermatological disease, skin damage or blemishes.
* Have participated in an investigational drug study within 30 days prior to screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keshava Kumar, PhD, MHSA, Study Director — Watson Laboratories
Locations (3):
- United States (3):
  - Watson investigational site, Miramar, Florida
  - Watson investigational site, Omaha, Nebraska
  - Watson investigational site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Transdermal Systems: Testosterone Transdermal System was applied daily starting at 4 mg, titratable to 6 mg or 2 mg based on testosterone serum concentration.
Period: Overall Study
Arm/Group | Testosterone Transdermal Systems
Started | 40
Baseline Characteristics Measured | 35
Completed | 35
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — did not meet inclusion criteria | 4

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone Transdermal Systems
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Time-average (Cavg) Steady State Testosterone Concentration Over 24 Hours
Description: A 24-hour pharmacokinetic sampling was performed on Day 28/29 after the start of dosing.
Time Frame: Day 28/29
Population: Per-protocol Population was used for the analysis. PP population included subjects who completed the treatment period of the study, who did not have more than two consecutive missing data, and who did not have any major protocol deviations.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Transdermal Systems
Number analyzed (Participants) | 35
ng/dL | 463 (122.1)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Testosterone Transdermal Systems
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 9/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Transdermal Systems (N=40)
Application site pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Application site vesicles (Skin and subcutaneous tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less